CLINICAL TRIAL: NCT01153152
Title: Study of Pain Following Removal of Wisdom Teeth With Acute Pulpitis
Status: Completed | Type: Observational
Sponsor: Wuhan University (Other)
Other Study IDs: NO.2009128
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2009-02

CONDITIONS: Pain
Keywords: wisdom teeth; acute pulpitis; extraction; pain; Pain Following Removal of Wisdom Teeth with Acute Pulpitis
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether pulp chamber opening and drainage on wisdom teeth with acute pulpitis before the extraction could reduce postoperative pain so beneficial to patient.

ELIGIBILITY:
Inclusion Criteria:

* inclusion criteria of upper wisdom teeth for the two groups were: vertical eruption; being worthless to be restored; deep caries in the occlusion surface with acute pain; without caries or acute pulpitis in the adjacent second molar

Exclusion Criteria:

* systemic diseases, smokers, inflammation in oral cavity,with history of psychiatric illness,pregnant or lactating females

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients requiring surgical removal of a single upper wisdom tooth with acute pulpitis were included in this prospective study
Sampling Method: Probability Sample
Dates: Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- School and Hospital of Stomatology, Wuhan University, Wuhan, Hubei, China